CLINICAL TRIAL: NCT07286305
Title: Media and Mental Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00005488
Record Dates: First submitted 2025-12-10; First posted 2025-12-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Mental and Behavioral Disorders; Mental Resilience; Emotional Awareness; Emotional Development
Keywords: Healthy Adults; Emotional Awareness
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into either a control group (media only), or an interventional group (ThinkHuman TV). There is a 50/50 chance of being assigned to each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Media Only (No Intervention)
- ThinkHuman TV (Active Comparator)
  Interventions: Device: ThinkHumanTV

INTERVENTIONS:
Device: ThinkHumanTV — Emotional Education Program
  Arms: ThinkHuman TV

SUMMARY:
This study's goal is to find if using the ThinkHumanTV program during 6 weekly sessions of watching Netflix or Disney series or movies for 90 minutes, together with 4 - 8 members of the Whole Health Center and EpiCenter and a discussion leader, improves the wellbeing of the group participants.

DETAILED DESCRIPTION:
This study's goal is to find out whether 6 weekly sessions of watching certain TV series or movies in a group setting, augmented through education from ThinkHuman TV about emotions and coping with emotions embedded in the process of watching (with a discussion leader), will improve the resilience of mental health patients enrolled in a long-term community mental health center. This will be tested by comparing ThinkHuman TV augmented movies with watching moving in a group without ThinkHuman TV educational activities to see if there is better improvement in resilience and well-being of the group participants who have THinkHuman included as compared to those who do not.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18years old
2. Recipient of treatment at WHC for at least 6 months.
3. English speaking

Exclusion Criteria:

1. Actively manic
2. Actively suicidal
3. Has not been dependent on drugs or alcohol for at least 30 days
4. Deemed to be at significant risk of being dangerous to self or others by the patients' WHC physician
5. Deemed inappropriate based on judgment of WHC physician informed by WHC staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-02-06 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in emotional awareness/intelligence. | 3 month interventional period
  Assessed using The Emotional Regulation Questionnaire
  * Score: Minimum = 0 Maximum = 70 (higher better outcome) Assessed using Emotional Self-Efficacy Scale
  * Score: Minimum = 32 Maximum = 160 (higher better outcome)
Change from baseline in anxiety. | 3 month interventional period
  Assessed using The Overall Anxiety Severity and Impairment Scale (OASIS)
  -Score: Minimum = 0 Maximum = 20 (higher worse outcome)
Change from baseline in depression symptoms. | 3 month interventional period
  Assessed using the Center for Epidemiologic Studies Depression scale (CES-D)
  -Score: Minimum = 0 Maximum = 30 (higher worse outcome)

SECONDARY OUTCOMES:
Change from baseline in quality of life. | After 3 month interventional period
  Assessed by Q-LES-Q-SF questionnaire
  -Score: Minimum = 14 Maximum = 70 (higher better outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
A limited data set (including all study data with identifiers other than date removed) will be shared by secure file transfer to consultants at Affectifi, Inc and will be available by request from the study investigators upon request through secure file transfer.
  Only general summary information will be shared with the study funder.